CLINICAL TRIAL: NCT02686892
Title: An Epidemiological Study of the Incidence of Inflammatory Bowel Disease in Spain
Acronym: INCIDENCIA
Status: Completed | Type: Observational
Sponsor: Javier P. Gisbert (Other)
Collaborators: Grupo Español de trabajo en Enfermedad de Crohn y Colitis Ulcerosa (GETECCU) (Unknown)
Responsible Party: Sponsor-Investigator, Javier P. Gisbert, MD PhD, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Other Study IDs: GIS-2015-INCIDENCIA
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2021-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflamatory bowel disease; Crohns disease; ulcerative colitis; incidence; epidemiology
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group: Spanish territory population of 46,439,864 inhabitants
- Cohort: Incident cases diagnosed with IBD over 12 months in the Spanish territory

SUMMARY:
This is a prospective, observational, multicenter, population-based incidence cohort study which will enroll cases of IBD (CD, UC, or indeterminate colitis) diagnosed in adults over 1 year in Spain.

In addition, each incident case that gave his/her informed consent, will be followed up for 12 months to determine changes in phenotype or disease location, the need for immunosuppressive and biologic treatments, and the need for hospital admissions and surgery during the first year after diagnosis.

DETAILED DESCRIPTION:
Study design This is a prospective, observational, multicenter, population-based incidence cohort study which will enroll cases of IBD (CD, UC, or indeterminate colitis) diagnosed in adults over 1 year in Spain.

In addition, each incident case that gave his/her informed consent, will be followed up for 12 months to determine changes in phenotype or disease location, the need for immunosuppressive and biologic treatments, and the need for hospital admissions and surgery during the first year after diagnosis.

Study population Incident cases diagnosed with IBD over 12 months in the Spanish territory, which has a population of 46,439,864 inhabitants (1 January 2015) according to data from the National Statistics Institute (INE). According to recent data, only 3% of incident cases are diagnosed in the pediatric population, so the study will focus on adult patients (over 15 years of age).

Case detection In Spain, health care is performed mostly by the public health services. According to recent data, approximately 15% of the Spanish population has private health insurance (Informe Sanidad Privada: Aportando Valor. Análisis de situación 2014 (Report on Private Health Care: Providing Value. 2014 Situation Analysis); available at: https://www.fundacionidis.com/wp-content/informes/informe_analisis situac_2014_0.pdf). In addition, of those persons having private health insurance, only about 15% make exclusive use of it. For these reasons and taking into account the specific characteristics of IBD, the risk of underestimating the incidence of IBD considering only cases seen in public health centers would be of little relevance. Therefore, this study will be conducted at centers providing public health care within the National Health System.

Furthermore, as previously mentioned, according to recent data only 3% of incident cases are diagnosed in the pediatric population, so the study will focus on adult patients (over 16 years of age)4.

To conduct this research project, an IBD specialist who is a member of GETECCU has been selected from each Autonomous Community, who will act as the coordinator in their region. Gastroenterologists in charge of IBD Units in Spain will be contacted, or if unavailable, a gastroenterologist from each of the hospitals included in the National Catalog of Hospitals as of 31 December 2014 at http://www.msssi.gob.es/ciudadanos/prestaciones/centrosServiciosSNS/hospitales/ home.htm (last accessed 13 August 2015). The most appropriate strategy for identification of cases will be planned on a case by case basis in each Autonomous Community, according to the specific characteristics of this Community, each province and health area, with the aim of detecting all incident cases. The databases of the endoscopy units and pathology departments will be reviewed in all sites participating in the study during the year of enrollment, in order to detect any possible incident cases of IBD that not might not have been identified initially.

Each participating investigator will confirm the diagnosis at the time of entering patients in the study and 3 months later to assure this diagnosis and the phenotypic characteristics of the disease, and thereby have greater diagnostic accuracy. External monitoring of incident cases included in the registry will also be performed by review of cases selected at random by the research team of Hospital Universitario de la Princesa.

Health areas in which detection and enrollment of all incident cases cannot finally be assured will be excluded from the study.

Definitions

* Disease location and phenotype: IBD location and phenotype will be defined according to the Montreal classification.
* Time to diagnosis: It will be defined as the time from the first medical consultation made by the patient after onset of symptoms to the diagnosis of IBD.
* Population center: The type of population center at the patient's birth and at diagnosis of IBD will be recorded. Whether the population center of origin of the patient is considered rural or urban will be based on the classification of the National Statistics Institute (INE) of each municipality.
* Socioeconomic level: Socioeconomic level will be assessed through different variables, such as the patient's educational level (primary education or lower, secondary education, higher education or equivalent), occupational status (self-employed, employee, unemployed, retired), professional status (nonsalaried or salaried) and type of working hours (full time or part time).
* Number of cohabitants: The number of cohabitants in the patient's home during childhood (up to 16 years) and at diagnosis of IBD will be recorded.
* Smoking: Smoking status will be categorized as "nonsmoker", "smoker", or "ex-smoker", and will be considered at the time of diagnosis of IBD. Patients will be considered "smokers" if they have a smoked more than 7 cigarettes per week for at least 6 months or smoked at least 1 cigarette in the 6 months prior to diagnosis. Patients will be considered "ex-smokers" l if they quit smoking at least 6 months before diagnosis. Patients will be considered "nonsmokers" if they never smoked or did so in a very small amount or occasionally.
* Treatments: Treatments received by the patient in the 12 months since diagnosis of the disease will be included, provided they were received for IBD. Only the first prescription of each therapeutic group will be recorded.
* Changes in phenotype: Changes in phenotype will be considered as the appearance of new lesions not present at diagnosis subsequent to the initial tests performed to determine disease extent and severity. In these cases, the phenotype, the complication leading to classification of the patient in a different phenotype and date of occurrence of the complication will be recorded.
* Hospital admission Hospital admission occurring during the first year from diagnosis of the disease will be included. The date of admission, date of discharge, if related or not to IBD and the cause of admission.
* Surgical procedures: The surgical procedures performed on the patient since diagnosis of IBD (including those performed before knowing the patient had IBD and which led to its diagnosis), the indication for surgery and the date of surgery will be recorded. An emergency surgical procedure will be considered as any surgery performed within 24 from admission of the patient to the emergency department. An elective surgical procedure will be considered as any procedure performed subsequent to the first day of admission and by the usual surgical team.

Data collection and follow-up:

Demographic data (age, sex, smoking), family history of IBD, socioeconomic characteristics, IBD type, pattern, and location and presence of extraintestinal manifestations at diagnosis will collected from each patient. The occurrence of complications (fistulas, stenosis, abscesses), changes in disease location, treatments for IBD, surgeries for IBD, and hospital admission during the first year since diagnosis will also be recorded.

After the patient is included, two other visits will be recorded during the 12 months, coinciding with the routine visits of the patient for follow-up of his/her disease. Thus, over the course of the study, 3 visits will be recorded, as described below:

* Visit 0 (baseline): inclusion of patient in the study and collection of socioeconomic data and on diagnosis of IBD.
* Visit 1 (month 3): confirmation of IBD diagnosis and updating of data related to treatment, changes in phenotype, hospital admissions, and surgery.
* Visit 2 (month 12): confirmation of IBD diagnosis and updating of data related to treatment, changes in phenotype, hospital admissions, and surgery. End of study.

In the case of patients not included at the time of diagnosis or later because they were referred from other centers, the corresponding visits will be performed retrospectively, completing the data retrospectively in the other visits (the previous ones). In addition, the inclusion period will be extended for 6 months in which patients diagnosed during the year of the study belonging to a participating area and not previously identified by the responsible investigator may be enrolled.

In the case of sites participating in ENEIDA, to avoid duplication of recording of the data by the responsible physician, the possibility of modifying the database will be proposed to the ENEIDA committee, including, in such a way that they are only visible to the investigators of this research project, the necessary variables that are not included in ENEIDA. In the event that this modification is not accepted by the ENEIDA committee, the study data will be recorded in an electronic database created specifically for this purpose.

In any case, the sites not currently participating in ENEIDA will record the data in an electronic database of REDCap created for this purpose. Subsequently, the two databases, both ENEIDA and that created specifically for the study, can be exported and combined for their analysis.

Statistical analysis The reference population for the study will be made up of the reference population of the areas of the public centers where the participating study physicians work, which will be based on the estimates of the National Statistics Institute (INE). The incidence rate (number of incident cases per 100,000 inhabitants) during 1 year will be calculated. Age-standardized incidence rates adjusted to the European population will be calculated6.

For qualitative variables, percentages will be calculated (with their 95% confidence intervals) and for quantitative variables, the arithmetic mean and standard deviation will be determined. In the univariate analysis, categorical variables will be compared using a Chi-squared (X2) test and quantitative variables will be compared using the appropriate test (Student's t-test, Wilcoxon, etc. depending on whether their values follow a normal distribution or not). To examine in detail the time course of the use of treatments, hospital admissions, surgery or occurrence of complications, the Kaplan-Meier method will be used, and the differences between the curves will be compared with the log-rank test. A Cox regression model will be used to study which variables are associated with the probability of occurrence of complications, progression to more severe phenotypes, use of immunosuppressive or biologic drugs, hospital admission, and performance of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age diagnosed with IBD.
* Diagnosis of IBD according to European Crohns and Colitis Organisation (ECCO) criteria.
* The patient must belong to the health area of one of the participating center

Exclusion Criteria:

* Patients who do not accept to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive observational study in which the whole Spanish population will be considered and which will include all incident cases of inflammatory bowel disease occurring in a year.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2017-01; Primary Completion 2019-02 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with the incidence of inflammatory bowel disease in Spain | 1 year

SECONDARY OUTCOMES:
Number of patients with incidece of inflammatory bowel disease in diferent regions of the spanish territory | 1 year
Characteristics of patients at diagnosis of inflammatory bowel disease | 1 year
  Type of IBD, extension of the IBD, severity of the IBD at diagnosis
Resourses used in the first year after diagnosis. | 1 year
  immunosuppressive treatments, biologic drugs, surgery, and hospital admissions
Delay from onset of symptoms to diagnosis of the disease | 1 year
  start date of symptoms, date of first visit to the family doctor, date of first visit to specialist, date of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Javier P Gisbert, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (16):
- Spain (16):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Clínico Universitario 'Lozano Blesa', Zaragoza, Aragon
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Gran Canaria Dr Negrín, Las Palmas, Canary Islands
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Hospital General de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital San Pedro de Alcántara, Cáceres, Extremadura
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital San Pedro, Logroño, La Rioja
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Galdakao -Usansolo, Usansolo, Vizcaya
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Shivananda S, Lennard-Jones J, Logan R, Fear N, Price A, Carpenter L, van Blankenstein M. Incidence of inflammatory bowel disease across Europe: is there a difference between north and south? Results of the European Collaborative Study on Inflammatory Bowel Disease (EC-IBD). Gut. 1996 Nov;39(5):690-7. doi: 10.1136/gut.39.5.690. PMID 9014768
- [Background] Kim HJ, Hann HJ, Hong SN, Kim KH, Ahn IM, Song JY, Lee SH, Ahn HS. Incidence and natural course of inflammatory bowel disease in Korea, 2006-2012: a nationwide population-based study. Inflamm Bowel Dis. 2015 Mar;21(3):623-30. doi: 10.1097/MIB.0000000000000313. PMID 25647154
- [Background] Burisch J, Pedersen N, Cukovic-Cavka S, Brinar M, Kaimakliotis I, Duricova D, Shonova O, Vind I, Avnstrom S, Thorsgaard N, Andersen V, Krabbe S, Dahlerup JF, Salupere R, Nielsen KR, Olsen J, Manninen P, Collin P, Tsianos EV, Katsanos KH, Ladefoged K, Lakatos L, Bjornsson E, Ragnarsson G, Bailey Y, Odes S, Schwartz D, Martinato M, Lupinacci G, Milla M, De Padova A, D'Inca R, Beltrami M, Kupcinskas L, Kiudelis G, Turcan S, Tighineanu O, Mihu I, Magro F, Barros LF, Goldis A, Lazar D, Belousova E, Nikulina I, Hernandez V, Martinez-Ares D, Almer S, Zhulina Y, Halfvarson J, Arebi N, Sebastian S, Lakatos PL, Langholz E, Munkholm P; EpiCom-group. East-West gradient in the incidence of inflammatory bowel disease in Europe: the ECCO-EpiCom inception cohort. Gut. 2014 Apr;63(4):588-97. doi: 10.1136/gutjnl-2013-304636. Epub 2013 Apr 20. PMID 23604131
- [Background] Niewiadomski O, Studd C, Hair C, Wilson J, McNeill J, Knight R, Prewett E, Dabkowski P, Dowling D, Alexander S, Allen B, Tacey M, Connell W, Desmond P, Bell S. Health Care Cost Analysis in a Population-based Inception Cohort of Inflammatory Bowel Disease Patients in the First Year of Diagnosis. J Crohns Colitis. 2015 Nov;9(11):988-96. doi: 10.1093/ecco-jcc/jjv117. Epub 2015 Jun 30. PMID 26129692
- [Background] Fernandez A, Hernandez V, Martinez-Ares D, Sanroman L, de Castro ML, Pineda JR, Carmona A, Gonzalez-Portela C, Salgado C, Martinez-Cadilla J, Pereira S, Garcia-Burriel JI, Vazquez S, Rodriguez-Prada I; EpiCom Group. Incidence and phenotype at diagnosis of inflammatory bowel disease. Results in Spain of the EpiCom study. Gastroenterol Hepatol. 2015 Nov;38(9):534-40. doi: 10.1016/j.gastrohep.2015.03.001. Epub 2015 Apr 15. PMID 25890448
- [Background] Lucendo AJ, Hervias D, Roncero O, Lorente R, Bouhmidi A, Angueira T, Verdejo C, Saluena I, Gonzalez-Castillo S, Arias A. Epidemiology and temporal trends (2000-2012) of inflammatory bowel disease in adult patients in a central region of Spain. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1399-407. doi: 10.1097/MEG.0000000000000226. PMID 25341061
- [Background] Anton Martinez J, Ortega Gomez A, Arranz Carrero A, Molina Sanchez A, Alvarez Garcia JF, Moreiras Jimenez JL, Gonzalez Blanco P, Gutierrez Sampedro N, Torres Garcia E. [Incidence of inflammatory bowel disease in the health area of Navalmoral de la Mata (Caceres, Spain) between 2000 and 2009]. Gastroenterol Hepatol. 2010 Dec;33(10):694-9. doi: 10.1016/j.gastrohep.2010.08.004. Epub 2010 Nov 3. Spanish. PMID 21051113
- [Background] Lopez-Serrano P, Perez-Calle JL, Carrera-Alonso E, Perez-Fernandez T, Rodriguez-Caravaca G, Boixeda-de-Miguel D, Fernandez-Rodriguez CM. Epidemiologic study on the current incidence of inflammatory bowel disease in Madrid. Rev Esp Enferm Dig. 2009 Nov;101(11):768-72. doi: 10.4321/s1130-01082009001100004. PMID 20001154
- [Background] Arin Letamendia A, Burusco Paternain MJ, Borda Celaya F, Pueyo Royo A, Martinez Echeverria A, Jimenez Perez FJ. Epidemiological aspects of inflammatory bowel disease in the Pamplona area. Rev Esp Enferm Dig. 1999 Nov;91(11):769-76. English, Spanish. PMID 10601770
- [Background] Rodrigo L, Riestra S, Nino P, Cadahia V, Tojo R, Fuentes D, Moreno M, Gonzalez Ballina E, Fernandez E. A population-based study on the incidence of inflammatory bowel disease in Oviedo (Northern Spain). Rev Esp Enferm Dig. 2004 May;96(5):296-305. doi: 10.4321/s1130-01082004000500002. English, Spanish. PMID 15180441
- [Background] Garrido A, Martinez MJ, Ortega JA, Lobato A, Rodriguez MJ, Guerrero FJ. Epidemiology of chronic inflammatory bowel disease in the Northern area of Huelva. Rev Esp Enferm Dig. 2004 Oct;96(10):687-91; 691-4. doi: 10.4321/s1130-01082004001000003. English, Spanish. PMID 15537375
- [Background] Saro Gismera C, Lacort Fernandez M, Arguelles Fernandez G, Anton Magarzo J, Garcia Lopez R, Navascues CA, Suarez Gonzalez A, Diaz Alvarez G, Gonzalez Bernal A, Palacios Galan A, Altadill Arregui A, Vizoso F. [Incidence and prevalence of inflammatory bowel disease in Gijon, Asturias, Spain]. Gastroenterol Hepatol. 2000 Aug-Sep;23(7):322-7. Spanish. PMID 11002532
- [Background] Lopez Miguel C, Sicilia B, Sierra E, Lopez Zaborras J, Arribas F, Gomollon F. [Incidence of inflammatory bowel disease in Aragon: outcome of a prospective population-based study]. Gastroenterol Hepatol. 1999 Aug-Sep;22(7):323-8. Spanish. PMID 10535203
- [Background] Monferrer Guardiola R, Martin Jimenez JA, Pedraza Sanz RG, Moreno Sanchez I, Soler Bahilo E, Hinojosa del Val J. Incidence of inflammatory bowel disease in the 02 health area of Castellon (1992-1996). Rev Esp Enferm Dig. 1999 Jan;91(1):33-46. English, Spanish. PMID 10089786
- [Background] Brullet E, Bonfill X, Urrutia G, Ruiz Ochoa V, Cueto M, Clofent J, Martinez Salmeron JF, Riera J, Obrador A. [Epidemiological study on the incidence of inflammatory bowel disease in 4 Spanish areas. Spanish Group on the Epidemiological Study of Inflammatory Bowel Disease]. Med Clin (Barc). 1998 May 16;110(17):651-6. Spanish. PMID 9656209
- [Background] Cella Lanau J, Lopez Zaborras J, Gomollon Garcia F, Sainz Samitier R. [Inflammatoru bowel disease in Aragon: a more and more frequent diagnosis]. Rev Esp Enferm Dig. 1995 May;87(5):363-7. Spanish. PMID 7626295
- [Background] Mate-Jimenez J, Munoz S, Vicent D, Pajares JM. Incidence and prevalence of ulcerative colitis and Crohn's disease in urban and rural areas of Spain from 1981 to 1988. J Clin Gastroenterol. 1994 Jan;18(1):27-31. doi: 10.1097/00004836-199401000-00008. PMID 8113581
- [Background] Martinez-Salmeron JF, Rodrigo M, de Teresa J, Nogueras F, Garcia-Montero M, de Sola C, Salmeron J, Caballero M. Epidemiology of inflammatory bowel disease in the Province of Granada, Spain: a retrospective study from 1979 to 1988. Gut. 1993 Sep;34(9):1207-9. doi: 10.1136/gut.34.9.1207. PMID 8406155
- [Background] Sola Lamoglia R, Garcia-Puges AM, Mones Xiol J, Badosa Gallart C, Badosa Gallart J, Casellas F, Pujol Pi J, Varea V. [Chronic inflammatory intestinal disease in Catalonia (Barcelona and Gerona)]. Rev Esp Enferm Dig. 1992 Jan;81(1):7-14. Spanish. PMID 1547040
- [Background] Alonso P, Ulla M, Soriano M, Aquise M, Del Villar V. [Intestinal inflammatory disease in the province of Soria. Retrospective clinical and epidemiologic study from 1981 to 1990]. Rev Esp Enferm Dig. 1992 Aug;82(2):87-91. Spanish. PMID 1389554
- [Background] Brullet E, Rue M, Montserrat A, Gil M, Malet A, Mas P, Bonfill X. [A descriptive epidemiological study of ulcerative colitis in a community hospital (1985-1989)]. Med Clin (Barc). 1991 Jun 8;97(2):45-9. Spanish. PMID 1895781
- [Background] Hinojosa J, Primo J, Lledo S, Lopez A, Roig JV, Fernandez J. [Incidence of inflammatory bowel disease in Sagunto]. Rev Esp Enferm Dig. 1990 Nov;78(5):283-7. Spanish. PMID 2090171
- [Background] Ruiz V. Crohn's disease in Galicia, Spain. Scand J Gastroenterol Suppl. 1989;170:29-31; discussion 50-5. doi: 10.3109/00365528909091346. PMID 2617188
- [Background] Sebastian Domingo JJ, Banares Canizares R, Velo Bellver JL, Clemente Ricote G, Cos Arregui E. [The epidemiological aspects of chronic inflammatory intestinal disease in a catchment area of the Autonomous Community of Madrid]. An Med Interna. 1989 Oct;6(10):519-22. Spanish. PMID 2491045
- [Background] Pajares Garcia JM, Rodriguez Munoz S, Mate Jimenez J. [Prevalence of Crohn disease in the central zone of Spain (Castillas, La Mancha, Cantabria and Rioja): cooperative epidemiologic study of the Castilian Digestive System Association]. Rev Esp Enferm Apar Dig. 1987 Apr;71(4):313-7. No abstract available. Spanish. PMID 3602564
- [Background] Ruiz Ochoa V. [Epidemiologic study of Crohn's disease in Galicia from 1976 to 1983]. Rev Esp Enferm Apar Dig. 1984 Oct;66(4):273-9. No abstract available. Spanish. PMID 6515083
- [Background] Martinez G, Fernandez Y, Rodrigo Saez L, Martinez E. [Epidemiologic study of Crohn's disease in the Asturian region]. Rev Esp Enferm Apar Dig. 1983 Jun;63(6):534-41. No abstract available. Spanish. PMID 6878842